CLINICAL TRIAL: NCT06934486
Title: A Multi-Centre Prospective, Non-Comparative, Open, Post-Marketing Surveillance Study to Obtain Clinical Outcome Data on the Use of Tissue Patch in the Prevention of Air Leaks Following Lung Resection
Brief Title: Observational Study of TissuePatch SF in Prevention of Air Leaks Following Lung Resection
Status: Not yet recruiting | Type: Observational
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Other Study IDs: SUR-25TP001
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Post-operative Air Leaks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with intra-operative air leak detected during lung resection
  Interventions: Device: TissuePatch Sealant Film

INTERVENTIONS:
Device: TissuePatch Sealant Film — Sealant film

SUMMARY:
Post-market, observational study to assess effectiveness of TissuePatch SF in managing/preventing air leaks after lung resection.

DETAILED DESCRIPTION:
Post-market study conducted to assess the continuing effectiveness and safety of TissuePatch SF when used as an adjunct to standard suture/staple closure of clinically significant (Macchiarini Grade ≥1) intra-operative visceral pleural air leaks incurred during lobectomy and segmentectomy (open or minimally invasive), including those performed as video-assisted thoracic surgery (VATS), in adults.

ELIGIBILITY:
Inclusion Criteria:

1. Is ≥18 and <80 years of age
2. Undergoing planned (not emergent) video-assisted thoracic surgery pulmonary resection
3. Understands and is willing to comply with all study related procedures
4. Has provided signed informed consent

Exclusion Criteria:

1. Women who are pregnant or lactating or, if of childbearing potential, are unwilling to use birth control for 6-months following surgery
2. Has severe congestive heart failure, pulmonary or renal failure, serious haematological disorder or significant liver disease
3. Has previously undergone a pneumonectomy
4. Has a bronchial fistula
5. Has or is suspected of having an active infection at or near the planned surgical site
6. Has a known allergy or sensitization to TissuePatch SF or its constituent components
7. In the investigator's opinion, has a life expectancy of less than 12 months
8. Has, in the investigator's opinion, any disease or condition, physical or psychological, that could interfere with the evaluation of TissuePatch SF or compliance with study procedures

Intra-Operative Exclusion Criteria:

1. >3 identified air leaks
2. No air leaks Macchiarini Grade ≥1

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing lung resection
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Intra-operative air leaks | Prior to the completion of surgery
  Air leaks successfully sealed or reduced as assessed by a submersion air leak test

SECONDARY OUTCOMES:
Overall device safety | 3-months post surgery
  Incidence of serious adverse events
Overall device safety | 6-months post-surgery
  Adverse events probably or causally related to the study device

IPD SHARING:
Plan to Share IPD: No